CLINICAL TRIAL: NCT03964038
Title: A Phase 1 Parallel Study to Assess the Relative Bioavailability of Gilteritinib Following a Single Dose of Gilteritinib Mini-tablet Oral Suspension and Gilteritinib Mini-tablets Compared to a Single Dose of Gilteritinib Tablet in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Gilteritinib Following a Single Dose of Gilteritinib Mini-tablet Oral Suspension and Gilteritinib Mini-tablets Compared to a Single Dose of Gilteritinib Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0602
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteer
Keywords: gilteritinib; ASP2215; Healthy volunteer
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- gilteritinib (Active Comparator): Participants will receive a single dose of gilteritinib under fasting conditions.
  Interventions: Drug: gilteritinib
- gilteritinib mini-tablet oral suspension (Experimental): Participants will receive a single dose of gilteritinib oral suspension with water under fasting conditions.
  Interventions: Drug: gilteritinib mini tablet
- gilteritinib mini-tablet (Experimental): Participants will receive a single dose of gilteritinib mini-tablets under fasting conditions.
  Interventions: Drug: gilteritinib mini tablet

INTERVENTIONS:
Drug: gilteritinib — oral
  Other Names: ASP2215
  Arms: gilteritinib
Drug: gilteritinib mini tablet — oral
  Other Names: ASP2215
  Arms: gilteritinib mini-tablet; gilteritinib mini-tablet oral suspension

SUMMARY:
The purpose of this study is to assess the relative bioavailability as well as the safety and tolerability of single doses of gilteritinib mini-tablets oral suspension and gilteritinib mini tablets compared to gilteritinib tablets under fasting conditions in healthy male and female participants.

DETAILED DESCRIPTION:
Participants will be screened for up to 28 days prior to investigational product (IP) administration on day 1. Eligible participants will be admitted to the clinical unit on day -1 and will be residential for 10 days/9 nights.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 to 32.0 kg/m2, inclusive and weighs at least 50 kg at screening.
* Female subject is not pregnant and the following condition applies:

  * Subject is not a woman of childbearing potential.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 120 days after study treatment administration.
* Male subject must not donate sperm during the treatment period and for 120 days after study treatment administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 120 days after study treatment administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to gilteritinib, or any components of the formulations used.
* Subject has had previous exposure with gilteritinib.
* Subject has any of the liver function tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase and total bilirubin) ≥ 1.5 × upper limit of normal on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study treatment administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) interval of > 430 msec (for male subjects) and > 450 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease or a family history of long QT syndrome.
* Subject has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study treatment administration, except for occasional use of paracetamol (up to 2 g/day), topical dermatological products, including corticosteroid products and hormone replacement therapy (HRT).
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening.
* Subject has a history of consuming > 14 units for male subjects or 7 units for female subjects of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol at screening or on day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations or the clinical unit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of gilteritinib in plasma: area under the concentration-time curve from the time of dosing to 72 hours (AUC72) | Up to Day 9
  AUC72 will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of gilteritinib in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 9
  AUCinf will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of gilteritinib in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to Day 9
  AUClast will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of gilteritinib in plasma: maximum concentration (Cmax) | Up to Day 9
  Cmax will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to Day 18
  Adverse Events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered an investigational product (IP) and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Day 18
  Number of participants with potentially clinically significant laboratory values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to Day 18
  Number of participants with potentially clinically significant ECG values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to Day 18
  Number of participants with potentially clinically significant vital sign values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- EPCU - Parexel, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.